CLINICAL TRIAL: NCT05422131
Title: Collection of Capillary Fingerstick Blood, Venous Serum, and Venous K2EDTA Blood Samples From Subjects Receiving Clozapine Therapy
Brief Title: Clozapine Therapy Sample Collection - Method Comparison Study
Status: Completed | Type: Observational
Sponsor: Saladax Biomedical, Inc. (Industry)
Collaborators: Northwell Health (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Other Study IDs: SBI-CLZ-002
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Patients Prescribed Clozapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients Prescribed Clozapine
  Interventions: Device: MyCare Insite Clozapine Test

INTERVENTIONS:
Device: MyCare Insite Clozapine Test — The MyCare Insite Clozapine Test is a 2 reagent system designed to evaluate the level of antipsychotic drug clozapine in a patients blood using the near patient device the MyCare Insite Analyser.

SUMMARY:
The method comparison study involves capillary fingerstick blood, venous serum, and venous K2EDTA blood sample collection from human subjects receiving clozapine treatment and their clozapine concentration measurement using a validated mass spectrometry method, the automated immunoassay MyCare Psychiatry Clozapine Assay Kit manufactured by SBI, and the point of care MyCare Insite Clozapine Test manufactured by SBI. Clozapine measurements obtained using the MyCare Insite Clozapine Test are intended for investigational purposes only and shall not be used in the management of patients receiving clozapine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must meet all the following criteria to be eligible for enrollment into the study:

  1. Female or male subjects 21 years of age or older;
  2. Current treatment with clozapine with documentation of diagnosed psychiatric condition requiring treatment;
  3. Capable of understanding and complying with parameters as outlined in the protocol;
  4. Capable of understanding and providing written informed consent, approved by an Institutional Review Board (IRB) prior to the initiation of any screening or study specific procedures.

Exclusion Criteria:

* 1. Female or male subjects under the 21 years of age; 2. Unwilling or unable to follow protocol requirements or to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 150 unique subjects are required for the collection of at least 150 of each a capillary fingerstick blood, venous serum, and venous K2EDTA blood samples. A subset of at least 75 subjects will require two fingerstick blood samples. Subjects consisting of males and females, at least 21 years of age or older, who meet the protocol Inclusion / Exclusion criteria as described below.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Sample Analysis - Method Comparision | October, 2022
  Determine if the MyCare Insite Clozapine Test returns blood level results which are equivalent to results obtained using the MyCare Pyschiatry Assay Kit and LC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Robert Christenson, Principal Investigator — University of Maryland
Locations (1):
- Saladax Biomedical, Inc., Bethlehem, Pennsylvania, United States